CLINICAL TRIAL: NCT07028775
Title: Clinical Application Study and Evaluation of Clopidogrel Resistance-Related Biomarkers in Predicting the Recurrence of Ischemic Events After Cerebral Artery Stenting
Brief Title: Biomarkers of Clopidogrel Resistance for Predicting Ischemic Recurrence After Cerebral Artery Stenting
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20250425-08
Record Dates: First submitted 2025-05-21; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Cerebral artery stenting; Clopidogrel resistance; Biomarkers
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the clinical significance of clopidogrel resistance-associated biomarkers (TMAO, C1q, and C4BPα) in patients receiving cerebral artery stents, and to develop an integrated predictive model incorporating these novel biomarkers along with CYP2C19 genotyping data for accurate clopidogrel resistance prediction in Chinese populations. By establishing this multidimensional assessment system, we intend to provide reliable risk stratification for post-stenting ischemic events and in-stent restenosis, ultimately facilitating personalized antiplatelet therapy decisions in cerebrovascular interventions. The proposed model may serve as a valuable clinical tool to optimize treatment strategies and improve outcomes for stented patients at risk of clopidogrel resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, with ischemic stroke due to atherosclerotic cerebrovascular stenosis;
* Scheduled for cerebral artery stenting with standard dual antiplatelet therapy (aspirin 100 mg/day + clopidogrel 75 mg/day) for ≥3 months.

Exclusion Criteria:

* Cardioembolic stroke (e.g., with atrial fibrillation);
* Embolic stroke of undetermined source (ESUS);
* Perioperative stroke;
* Requiring intravenous thrombolysis (rt-PA, urokinase, alteplase, or tenecteplase);
* Mechanical thrombectomy;
* Current use of anticoagulants (warfarin, rivaroxaban, dabigatran, etc.);
* Severe hepatic or renal dysfunction;
* Allergy to clopidogrel or aspirin;
* Bleeding tendency (e.g., thrombocytopenia or active gastrointestinal ulcer);
* History of recurrent miscarriage or current pregnancy;
* Malignancy or life expectancy <1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from the inpatient department of neurology at Nanjing First Hospital.
Sampling Method: Probability Sample
Enrollment: 839 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Recurrent ischemic stroke | At 30 days, 90 days, 6 months, and 1 year after antiplatelet therapy
  Recurrent ischemic stroke is defined as either: 1) acute exacerbation of pre-existing deficits occurring ≥21 days post-initial event onset, or 2) emergence of novel neurological deficits (including transient ischemic attack and acute ischemic stroke). Diagnostic confirmation requires both clinical correlation with symptoms and neuroimaging evidence (MRI) demonstrating new cerebral infarction within the original vascular territory, or acute neurological symptoms (within 24 hours) localizing to the original vascular territory with absence of new cerebral infarction on MRI.

SECONDARY OUTCOMES:
In-stent restenosis | At 90 days after antiplatelet therapy
  Head-neck CTA

OTHER OUTCOMES:
ADP-induced platelet aggregation | At 72 hours and 30 days after antiplatelet therapy
  Whole blood platelet aggregation induced by ADP was detected by a whole-blood aggregometer (Chrono-Log model 590-2D, Chromo-Log Corp., Havertown, PA, USA). Changes in electronic resistance (Ω) values between two electrodes were recorded to reflect the rate of whole-blood platelet aggregation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No